CLINICAL TRIAL: NCT03206411
Title: Assessment of Severity and Outcome of Addicted Cases Admitted to Neurology and Psychiatry Hospital in Assiut University.
Brief Title: Assessment of Severity and Outcome of Addicted Cases.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sarah Abdelsamee Mohammed Ali, Principal Investigator, Assiut University
Other Study IDs: Addiction
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Addiction, Substance
MeSH Terms: conditions — Substance-Related Disorders | interventions — Liver Function Tests; Electrocardiography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Renal and liver function tests , ECG , Sex Hormones Profile — Renal Function tests as creatinine , Uric Acid , Blood urea. Liver Function tests as AST , ALT, ALP ECG (Electrocardiogram recording) SEX hormones as LH , FSH , and Testosterone

SUMMARY:
* Addiction to drugs and alcohol is increasingly becoming a worldwide trend that is prevalent in both rich and poor countries . Substance abuse shows a significant warming to the health, social and economic build of families, communities and nations. Extent of worldwide psychoactive substance use is estimated at 2 billion alcohol users and 185 million drug users .
* Substance abuse (including alcohol and drugs) is an important risk factor for poor health globally due to their intoxicating effects or their toxic effects on organs and tissues that lead to the development of diseases, injuries and other health conditions
* Drug abuse is associated with the increased risk of cardiovascular diseases. A study on the need for hospitalization in approximately 4800 drug users found that 223 of these were admitted to hospital due to cardiovascular diseases .
* The majority of abused substances or their metabolites are excreted through the kidneys and renal complications of drug abuse are very common .The involvement of the kidney due to drug abuse is either attributed to their elimination through the kidney, or a direct nephrotoxic effect. The damage may be acute and reversible, or chronic and can leads to end stage renal failure .
* Addiction is responsible for different types of liver diseases including fatty liver, hepatitis and liver failure. . Intravenous drug addiction by sharing of contaminated needle is very important risk factor for the development of liver diseases, particularly hepatitis B and hepatitis C. Globally, 90% of new hepatitis C infections are attributed to drug injection . In the long run, substance abuse has negative effects on sexual functions and leads to the onset of sexual disorders. .
* Long term use of alcohol was reported to inhibit of hypothalamic-pituitary-adrenal axis and reduces the release of gonadotropins from the pituitary . Morphine administration suppresses LH release and reduces the levels of testosterone, which affects testicular function.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are addicted for at least one year.

Exclusion Criteria:

* Patients who are addicted for less than one year.
* Patients with history of previous renal impairment
* Patients with history of hepatitis B, C or HIV infection
* Patients with history of autoimmune disease.
* Patients with history of heart disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are addicted for at least one year.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Sex Hormones Profile | 1 day
  Measure the changes in the Sex Hormones (LH , FSH and Testosterone) due to drug addiction in different people.

SECONDARY OUTCOMES:
Liver Function tests. | 1 day
  Measure the changes in the liver enzymes (AST,ALT and ALP) due to drug addiction in different people.
Renal Functions tests. | 1 day
  Measure the changes in the renal function due to drug addiction in different people.
ECG | 1 day
  Record the changes in the Electrocradiogram due to addiction

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No